CLINICAL TRIAL: NCT06852612
Title: Dietary Treatment Strategies and Metabolic Control in Glycogen Storage Disease Type I (GSD-DIET)
Brief Title: Dietary Treatment Strategies and Metabolic Control in Glycogen Storage Disease Type I
Acronym: GSD-DIET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Zurich (Other); University Hospital Freiburg (Other); University Hospital Heidelberg (Other); Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02154
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Glycogen Storage Disease Type I
Keywords: Gsd1; Metabolism; Fructose; Galactose
MeSH Terms: conditions — Glycogen Storage Disease Type I | interventions — Fructose; Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet with additional fructose intake (Experimental)
  Interventions: Dietary Supplement: Fructose
- Diet with additional fructose and galactose intake (Experimental)
  Interventions: Dietary Supplement: Fructose and galactose

INTERVENTIONS:
Dietary Supplement: Fructose — 40g fructose (free and bound, max amount of fructose from added free sugar/saccharose 25g)
  Arms: Diet with additional fructose intake
Dietary Supplement: Fructose and galactose — 10g galactose (mostly from lactose) plus 40g of fructose (free and bound, max amount of fructose from added free sugar/saccharose 25g)
  Arms: Diet with additional fructose and galactose intake

SUMMARY:
The present project will specifically assess metabolic effects of dietary interventions with controlled intake of fructose and fructose/galactose in GSDI, with the aim to provide evidence whether relaxed dietary restrictions of fructose and galactose may be justified in treatment recommendations at least for adults, which would considerably enlarge food choice in everyday life of the patients with an expected positive impact on the quality of life of patients with this rare disorder.

DETAILED DESCRIPTION:
To assess relaxed restriction of fructose and fructose/galactose intake on secondary metabolic alterations in GSDI, (i) by looking at the traditional parameters for assessing metabolic control in clinical chemistry (lactate, triglycerides, uric acid), and (ii) by using a broad analytical approach relying on targeted metabolomics/lipidomics.

It is hypothesized that relaxed restrictions on the intake of fructose and/or galactose as part of the diet in everyday life may lead to an increase in blood lactate levels (=primary outcome), triglycerides, and uric acid to a certain degree compared to baseline. However, this increase is expected to remain within a range that is not clinically relevant for adult patients, especially when fructose/galactose intake is not excessive and stays within the usual daily allowances for healthy individuals, as planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* Genetically and/or enzymatically confirmed diagnosis of GSDI (GSDIa or GSDIb)
* Male or female ≥ 18y
* Restriction of fructose intake in usual dietary treatment
* Written informed consent

Exclusion Criteria:

* Non-compliance with routine dietary treatment
* Pregnancy or lactation
* Liver transplant
* Recurrent hospitalisations due to metabolic decompensation within the last 12 months
* Severe chronic kidney disease with glomerular filtration rate (GFR) < 30 ml/min
* For GSDIb: Severe, uncontrolled symptomatic inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in lactate during the dietary intervention compared to baseline under the usual diet | 4 Weeks
  Lactate belongs to the parameters of secondary metabolic disturbance traditionally used to estimate metabolic control in GSDI in routine clinical practice (lactate, triglycerides, uric acid). Redundant measurements of lactate are performed in blood as well as in collected urine.

SECONDARY OUTCOMES:
Change in plasma triglycerides during the dietary intervention compared to baseline (as parameters traditionally measured together with lactate to estimate overall metabolic control) | 4 Weeks
Change in plasma uric acid during the dietary intervention compared to baseline (as parameters traditionally measured together with lactate to estimate overall metabolic control) | 4 Weeks
Plasma metabolite changes in targeted metabolomics during the dietary intervention compared to baseline measurements. | 4 Weeks
Plasma metabolite changes in targeted lipidomics during the dietary intervention compared to baseline measurements. | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michel Hochuli, MD, PhD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD will be made available starting 12 months after publication of trial results.
Access Criteria: Ethics approval, as applicable under Swiss legislation, will need to be obtained by those requesting the data. Additionally, a data transfer and processing agreement must be in place to ensure compliance with data protection regulations.